CLINICAL TRIAL: NCT01649479
Title: Comparative Prevalence of Psychiatric Manifestations in Purely Obstetrical Antiphospholipid Syndrome
Acronym: MENT-APL-O
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Impossible to include patients at a correct rate; patients don't want to come back so they refuse participation.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: PHRC-I/2012/FC-01; 2012-A00705-38 (Other: RCB number)
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Antiphospholipid Syndrome
Keywords: Obstetrical antiphospholipid syndrome; Thrombophilia
MeSH Terms: conditions — Antiphospholipid Syndrome; Thrombophilia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Suspected Obstetrical APS; confirmed APS (Other): The patients included in this study are women actively addressed to the participating departments because of clinical symptoms corresponding to suspected obstetrical anti-phospholipid syndrome.
  Bloodwork later confirms that these patients have APS.
  All patients included in this study will have the following interventions:
  * antiphospholipid antibody tests
  * thrombophilia bloodwork
  * psychiatric evaluation
  Interventions: Biological: Antiphospholipid antibody tests; Biological: Thrombophilia bloodwork; Other: Psychiatric evaluation
- Sus. Obst. APS, confirmed thrombophilia (Other): The patients included in this study are women actively addressed to the participating departments because of clinical symptoms corresponding to suspected obstetrical anti-phospholipid syndrome.
  Bloodwork later confirms that these patients are thrombophilic.
  All patients included in this study will have the following interventions:
  * antiphospholipid antibody tests
  * thrombophilia bloodwork
  * psychiatric evaluation
  Interventions: Biological: Antiphospholipid antibody tests; Biological: Thrombophilia bloodwork; Other: Psychiatric evaluation
- Suspected Obstectrical APS; unconfirmed (Other): The patients included in this study are women actively addressed to the participating departments because of clinical symptoms corresponding to suspected obstetrical anti-phospholipid syndrome.
  Bloodwork cannot confirm APS, nor thrombophilia.
  All patients included in this study will have the following interventions:
  * antiphospholipid antibody tests
  * thrombophilia bloodwork
  * psychiatric evaluation
  Interventions: Biological: Antiphospholipid antibody tests; Biological: Thrombophilia bloodwork; Other: Psychiatric evaluation

INTERVENTIONS:
Biological: Antiphospholipid antibody tests — Each patient will be tested for antiphospholipid antibodies.
Biological: Thrombophilia bloodwork — Bloodwork will be drawn up for:
  * antithrombin, protein C, protein S
  * Factor V Leiden polymorphisms (F5 1691A)
  * prothrombin 20210A gene polymorphism (F2 20210A)
  * JAK2 617F Mutation
  * Homocysteine
  * Factor VIII
Other: Psychiatric evaluation — During this consultation, the Mini International Neuropsychiatric Interview will be used to screen for psychiatric symptoms. Should the latter be detected, a further consult with a psychiatrist or a psychologist will be organized; this second consult will include the Mood Disorder Questionnaire (MDQ), the Beck Depression Inventory (BDI), the Inventory for Depressive Symptomatology - Clinician (IDS-C) and the Structured Clinical Interview for Disorders (SCID, DSM-IV).

SUMMARY:
The main objective of this study is to estimate the lifetime prevalence of major psychiatric disorders (axis I DSM-IV; Diagnostic and Statistical Manual of Mental Disorders, version IV) in a large sample of patients with developed clinical signs of pure obstetrical antiphospholipid syndrome (suspected APS).

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. To compare the lifetime prevalence of these major disorders between groups;

B. To assess the association of different, targeted, qualitative biomarkers with clinical symptomatology;

C. To assess the association between the presence of "transitory APS" and the presence of psychiatric disorders;

D. Estimate and compare the current prevalence (= the day of assessment) of major psychiatric disorders in the sample of patients who developed clinical signs of obstetrical APS;

E. Estimate the current prevalence (= the day of assessment) and intensity of major depressive episodes (MDE) in the sample of patients;

F. Compare the prevalence of current MDE and the intensity of depressive symptoms present between groups;

G. Estimate and compare the (lifetime and current) prevalence by category of psychiatric disorders (psychotic, anxiety, mood, etc..) in the APS group with that in the thrombophilic group and the remaining group;

H. To study the average age of onset of psychiatric disorders and clinical manifestations of APS in the sample of patients who developed clinical signs of obstetrical APS;

I. Compare the mean ages between groups;

J. Compare the mean age at onset of psychiatric disorders with the average age of the first clinical manifestation of the disease in the group of women with APS.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Not postmenopausal
* Able to understand the nature, purpose and methodology of the study and agreed to cooperate in clinical and biological assessments
* Available for 12 weeks of follow-up
* Isolated obstetric morbidity, defined by at least one of the following criteria:
* at least three consecutive episodes of unexplained, early, embryonic miscarriage, which occurred before the 10th week of pregnancy, with normal maternal anatomic and hormonal assessment, normal karyotypes for both biological parents;
* at least one unexplained fetal death, defined as occurring after the 10th week of pregnancy, involving a morphologically normal fetus as documented by ultrasound examination or direct examination of the conceptus;
* at least one premature birth of a morphologically normal fetus before the 34th week of pregnancy, because of: (1) pre-eclampsia, severe or not, according to the American College of Obstetrics and Gynecology, ACOG, 2002; (2)documented placental insufficiency, defined by the following parameters: (2a) abnormal or non-reassuring fetal monitoring exam, in general a non-reactive absence-of-fetal-stress test (fetal monitoring), suggesting fetal hypoxemia; (2b) a Doppler examination of uterine arteries suggesting fetal hypoxemia, ie the absence of end-diastolic flow in the umbilical arteries; (2c) oligohydramnios, that is to say, an amniotic flow index <5 cm; (2d) indexed birth weight for gestational age and sex below the 10th percentile.
* Patient willing to accept psychological and medical care over the long term

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient or breastfeeding
* Systemic vascular morbidity, defined by the following criteria: (1) Any personal history of venous thromboembolism, defined by the occurrence of deep phlebitis and / or a pulmonary embolism, diagnosed by means of objective exploration ; (2)Any personal history of superficial venous thrombosis; (3) Any personal history of clinical, symptomatic relapses of arterial insufficiency - the latter may be cerebro vascular in nature (transient ischemic attack, stroke, etc..), coronary in nature (angina, myocardial infarction, etc..) or otherwise (claudication mesenteric, etc.), and objectively diagnosed.
* Systemic inflammatory disease: any history of systemic disease, lupus erythematosus or other connective, rheumatoid arthritis
* Any history of neoplastic disease
* Chronic antithrombotic treatment taken before the occurrence of obstetrical complications
* Any chronic immunosuppressive therapy or immunomodulatory therapy (eg corticosteroids, hydroxochloroquine or intravenous immunoglobulins)
* Fetal loss can be explained by infectious, metabolic (including rates of fasting blood glucose> 7 mmol / L), anatomical or hormonal factors
* History of infection with hepatitis B, hepatitis C or HIV
* Taking antipsychotic treatment potentially implicated in biological autoimmune abnormalities

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
presence/absence of (lifetime) psychiatric symptoms | baseline (transversal); Day 0
  The Mini International Neuropsychiatric Interview (MINI 6) will be used to determined the presence/absence of (lifetime) psychiatric symptoms.

SECONDARY OUTCOMES:
presence/absence of (current) psychiatric symptoms | baseline (transversal); Day 0
  The Mini International Neuropsychiatric Interview (MINI 6) will be used to determined the presence/absence of (current) psychiatric symptoms.
SCID-1 score | baseline (transversal); Day 0 or up to Day 15
  Structured Clinical Interview for Disorders (SCID-1) score for patients with a positive MINI evaluation.
MDQ score | baseline (transversal); Day 0
  Mood Disorder Questionnaire score
BDI score | baseline (transversal); Day 0 or up to Day 15
  The Beck Depression Inventory (BDI) score for currently depressed patients only.
IDS-C score | baseline (transversal); Day 0 or up Day 15
  Inventory of Depressive Symptomatology (IDS-C) for currently depressed patients.
presence/absence of lupus anticoagulant | baseline (transversal); Day 0
presence/absence of anticardiolipid antibodies | baseline (transversal); Day 0
presence/absence of anti-beta2-glycoprotein 1 antibodies | baseline (transversal); Day 0
deficit in antithrombin: yes/no | baseline (transversal); Day 0
Deficit in protein C: yes/no | baseline (transversal); Day 0
Deficit in protein S: yes/no | baseline (transversal); Day 0
Excess of FVIII: yes/no | baseline (transversal); Day 0
  Excess of coagulation factor VIII?
Excess of homocystein? yes/no | baseline (transversal); Day 0
presence/absence of allele F5 1691A | baseline (transversal); Day 0
  F5 1691A: allele 1691A for the factor V leiden gene
presence/absence of allele F2 20210A | baseline (transversal); Day 0
  F2 20210A: allele 20210A for the prothrombin gene
presence/absence of allele JAK2 617F | baseline (transversal); Day 0
  JAK2 617F: 617f mutation at the jak2 gene
Age at beginning of psychiatric symptoms | baseline (transversal); Day 0
  in years
Age at beginning of APL or thrombophilia symptoms | baseline (transversal); Day 0
  in years

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - APHM - Hôpital de la Conception, Marseille
  - APHM - Hôpital La Timone Adultes, Marseille
  - APHM - Hôpital Nord, Marseille
  - CHU de Montpellier - Hôpital Saint-Eloi, Montpellier
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes